CLINICAL TRIAL: NCT02602704
Title: Effectiveness of Bazedoxifene for Prevention of Glucocorticoid-induced Bone Loss in RA Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanyang University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Yoon-Kyoung Sung, Associate professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUHRD-SPE-15-05; WI205578 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — bazedoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bazedoxifene & Calcium/Vit D (Active Comparator): * Enrollment: 57
  * Drug: Bazedoxifene 20 mg/day (Viviant)
  * Drug: Elemental calcium 1200mg daily and vitamin D 800 IU daily (Caltrate D 400 * 2/day)
  Interventions: Drug: Bazedoxifene; Drug: Calcium/Vit D
- Calcium/Vit D (Active Comparator): * Enrollment: 57
  * Drug: Elemental calcium 1200mg daily and vitamin D 800 IU daily (Caltrate D 400 * 2/day)
  Interventions: Drug: Calcium/Vit D

INTERVENTIONS:
Drug: Bazedoxifene — Bazedoxifene 20mg/day (Viviant) for 48 weeks
  Other Names: Viviant
  Arms: Bazedoxifene & Calcium/Vit D
Drug: Calcium/Vit D — Elemental calcium 1200mg daily and vitamin D 800 IU daily (Caltrate D 400 * 2/day) for 48 weeks
  Other Names: Hardcal Chewable

SUMMARY:
* The purpose of this study is to study the effectiveness of bazedoxifene in preventing loss of bone mineral density (BMD) and trabecular bone score (TBS), and any fractures in postmenopausal rheumatoid arthritis (RA) patients receiving long-term GCs.
* This is a randomized, controlled, open-label extension study for 48 or 56 weeks. At study entry, all patients will receive elemental calcium (1200 mg daily) and vitamin D (800 IU daily) and will be randomized by blocks of two to receive either bazedoxifene (20 mg/day) or none.

DETAILED DESCRIPTION:
* The purpose of this study is to study the effectiveness of bazedoxifene in preventing loss of bone mineral density (BMD) and trabecular bone score (TBS), and any fractures in postmenopausal rheumatoid arthritis (RA) patients receiving long-term GCs.
* This was a randomized, controlled, open-label study conducted for 56 weeks. Four trial visits occurred over the course of the 56 weeks. At study entry, all patients who took elemental calcium (1200 mg daily) and vitamin D (800 IU daily) were assigned by blocks of two to receive either bazedoxifene (20 mg/day) (bazedoxifene group) or not (control group).
* Randomization was performed by an independent coordinator. Participants were followed-up at 24 weeks and 48 weeks with special attention to RA flares and occurrence of AEs.
* Demographic characteristics such as age, sex, and medications related to RA, as well as laboratory result such as complete blood count (CBC), chemistry, and levels of inflammatory markers were collected at enrollment. BMD and trabecular bone score (TBS) were assessed at 0 and 48 weeks, and levels of bone turnover markers were assessed at 0, 24, and 48 weeks. At 56 weeks, the occurrence of AEs was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female RA patients ≥ 45 years old with self-reported postmenopausal for ≥12 months or prior hysterectomy with bilateral oophorectomy. Female patients ≥ 55 years old who had prior hysterectomy without oophorectomy or with unilateral oophorectomy.
* Having been receiving low to moderate dose of glucocorticoids (prednisone ≤7.5 mg/day or equivalent) for ≥3 months prior to entry. (When taking glucocorticoids PRN, prednisone ≥1mg/day in average.)
* Patients expected to be on glucocorticoid treatment for 3 months after entry.
* Patients with an osteopenic mean lumbar spine (LS; L1-L4) or femoral neck bone mineral density (BMD; -1 < T-score < -2.5)
* Patients who provide a written consent of participating in this study.

Exclusion Criteria:

* Patients with condition that may interfere with the evaluation of spinal or hip osteoporosis by DXA such as two or more vertebral (L1-L4) fractures or other vertebral deformity
* Patients with hypercoagulability risk factors or a history of deep vein thrombosis and pulmonary embolism
* History of allergic reactions or intolerance to bazedoxifene or other SERM
* Patients receiving bisphosphonates, parathyroid hormone, SERMs, or anticonvulsants therapies within 6 months prior to entry
* Patients with known bone disorders such as osteomalacia, renal osteodystrophy and hyperparathyroidism
* Patients with undiagnosed uterine bleeding
* Patients with severe renal impairment or creatinine clearance <30ml/min

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change of Bone Mineral Density (BMD) | Baseline and 48 weeks
  BMD of the L-spine (L1-4) and femur neck was assessed by dual-energy x-ray absorptiometry (DXA) (Hologic®, Discovery W, Hologic APEX software version 2.3.1; Bedford, MA, USA). BMD in the L-spine was estimated as the mean of individual measurements for L1-L4 excluding any fractured or otherwise deformed vertebrae. The technician who was responsible for measuring BMD was blinded to the details of the study.

SECONDARY OUTCOMES:
Change of Trabecular Bone Score (TBS) | Baseline and 48 weeks
  Lumbar spine TBS is obtained using the spine DXA scan archived from the baseline and 48 weeks tests. It is calculated after reanalysis of the DXA scan of the L-spine using TBS iNsight® software (Version 2.0.0.1, Med-Imaps, Bordeaux, France). Vertebrae excluded in the calculation of BMD are also excluded in the TBS calculation.
Development of the thoracic and lumbar vertebrae for deformities by visual inspection | Baseline and 48 weeks
  Baseline vertebral fracture is defined as a loss of at least 25% of vertebral height through the thoracic spine X-ray and the lumbar spine X-ray. Incident vertebral fractures at 48 weeks is diagnosed when there were distinct alterations in the morphology of the vertebral bodies that resulted in the loss of at least 25% of vertebral height of previously normal vertebrae.
  The location, the date of occurrence and the severity of fracture (mild, moderate, severe, etc.) are described.
Development of any fractures including nonvertebral fractures | Baseline, 24 weeks and 48 weeks
  Measured by the questionnaire for fracture. Check item: the location and the date of occurrence of fracture.
Change in serum C-terminal telopeptide (CTX) | Baseline, 24 weeks and 48 weeks
  Serum C-telopeptide levels (ng/ml) are assayed by electrochemiluminescence (Roche Diagnostics, GmbH, Mannheim, Germany). Blood samples are collected after at least an 8-hour fast.
Change in urine N-telopeptide (NTX) | Baseline, 24 weeks and 48 weeks
  Urine N-telopeptide levels (ng/ml) are measured by chemiluminescence (Ortho Clinical Diagnostics, New York, USA) using commercially available kits. Urine samples are collected after at least an 8-hour fast.
Change in serum bone specific alkaline phosphatase | Baseline, 24 weeks and 48 weeks
  Serum bone-specific alkaline phosphatase (ALP) levels (µg/L) are also determined by electrochemiluminescence using commercial kits (Beckman Coulter Inc., Brea, USA). Blood samples are collected after at least an 8-hour fast.
Change in serum osteocalcin | Baseline, 24 weeks and 48 weeks
  Serum osteocalcin levels (ng/mL) are also determined by electrochemiluminescence using commercial kits (Beckman Coulter Inc., Brea, USA). Blood samples are collected after at least an 8-hour fast.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Kyoung Sung, MD, PhD, MPH, Principal Investigator — Hanyang University Hospital for Rheumatic Diseases
Locations (1):
- Hanyang University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho SK, Song YJ, Kim HW, Nam E, Jeon JY, Yoo HJ, Sung YK. Comparative effectiveness of tofacitinib and tumour necrosis factor inhibitors in patients with rheumatoid arthritis in real-world practice: a prospective observational study. Rheumatology (Oxford). 2025 Feb 1;64(2):541-547. doi: 10.1093/rheumatology/keae109. PMID 38366621
- [Derived] Cho SK, Kim H, Lee J, Nam E, Lee S, Choi YY, Sung YK. Effectiveness of bazedoxifene in preventing glucocorticoid-induced bone loss in rheumatoid arthritis patients. Arthritis Res Ther. 2021 Jul 2;23(1):176. doi: 10.1186/s13075-021-02564-1. PMID 34215316